CLINICAL TRIAL: NCT05908630
Title: The Role of Accidental Hypothermia in Drowning-related Out-of-hospital Cardiac Arrest: A Danish Six-year Observational Cohort Study
Brief Title: Accidental Hypothermia in Drowning-related OHCA
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Niklas Breindahl, Medical Doctor, Prehospital Center, Region Zealand
Other Study IDs: DROWN_HYPOTHERMIA
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Hypothermia, Accidental; Hypothermia Due to Cold Environment; Drowning; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Hypothermia; Drowning; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normothermic drowning patients with OHCA.: First in-hospital temperature measurement (using any probe) within 6 hours after hospital admission ≥35C.
- Hypothermic drowning patients with OHCA.: First in-hospital temperature measurement (using any probe) within 6 hours after hospital admission <35C.
  Interventions: Other: Hypothermia

INTERVENTIONS:
Other: Hypothermia — Accidental hypothermia is defined as: "an involuntary drop in core body temperature <35C"
  Groups: Hypothermic drowning patients with OHCA.

SUMMARY:
This study aims to report mortality and neurological outcome 180 days after drowning incident in patients with accidental hypothermia vs normothermia following drowning-related OHCA in Denmark during a six-year period from 2016-2021.

DETAILED DESCRIPTION:
The incidence of accidental hypothermia in patients with out-of-hospital cardiac arrest (OHCA) due to drowning is prevalent. Accidental hypothermia is known to decrease oxygen consumption and hypoxic brain damage in patients with OHCA, but may result from prolonged submersion times, which is shown to increase drowning mortality and morbidity. However, many case reports present extraordinary instances of hypothermic patients with drowning-related OHCA surviving with a good neurological outcome despite prolonged submersion times. A larger, retrospective study is warranted to accurately investigate the role of accidental hypothermia in patients with drowning-related OHCA.

This study is a nationwide, retrospective cohort study with 180-days follow-up from 2016-2021 comparing survival and neurological outcome 180 days after drowning incident in normothermic (≥35C) vs hypothermic (<35C) patients with drowning-related OHCA. A total of 317 patients have been identified by the Danish Drowning Formula and manually validated (Breindahl et al, 2023, unpublished data). Prehospital data from the DCAR will be linked to in-hospital data using the patients' unique civil registration number and presented the "Utstein style". The primary outcome is composite of mortality or poor neurological outcome 180 days after drowning incident (modified Rankin Scale score > 3). Secondary outcomes include hospital length of stay (continuous), intensive care unit admission (binary) and length of stay (continuous), need for ECLS (binary) and duration (continuous), need for mechanical ventilation (binary) and duration (continuous), survival to hospital discharge, and 30-day survival.

The investigators expect to provide evidence on the role of accidental hypothermia in drowning-related OHCA to support evidence-based guidelines and improve clinical decision-making in the future.

ELIGIBILITY:
Inclusion Criteria - Drowning persons with:

* OHCA registered in the DCAR from 2016-2021.
* An in-hospital temperature measurement (using any probe) within 6 hours after hospital admission.

Exclusion Criteria - Drowning persons will be excluded if:

* They have obvious signs of irreversible death (decapitation, decomposition, post-mortem lividity, post-mortem rigidity).
* They are declared dead on scene.
* They have a valid Do-Not-Attempt-Resuscitation order or other code status orders limiting life-sustaining therapies.
* They do not have a valid civil registration number.
* They do not have a valid in-hospital temperature measurement (any probe within 6 hours after hospital admission).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Drowning persons with out-of-hospital cardiac arrest identified in the Danish Cardiac Arrest Registry (DCAR).
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Survival or poor neurological outcome | 180 days after drowning incident.
  The primary outcome is a composite of mortality or poor neurological outcome 180 days after drowning incident according to the Utstein style

SECONDARY OUTCOMES:
Hospital length of stay | Immediately after hospital discharge
  Continuous
Intensive care unit admission | Immediately after hospital discharge
  Binary
Intensive care unit length of stay | Immediately after hospital discharge
  Continuous
Need for ECLS | Immediately after hospital discharge
  Binary
Duration of ECLS | Immediately after hospital discharge
  Continuous
Need for mechanical ventilation | Immediately after hospital discharge
  Binary
Duration of mechanical ventilation | Immediately after hospital discharge
  Continuous
Survival to hospital discharge | Immediately after hospital discharge
  Binary
30-day survival | 30 days after drowning incident
  Binary

CONTACTS AND LOCATIONS:
Overall Officials: Helle Collatz Christensen, Study Director — Prehospital Center, Region Zealand
Locations (1):
- Prehospital Center, Næstved, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No